CLINICAL TRIAL: NCT02824081
Title: Neuroinflammation, Serotonin, Impulsivity and Suicide
Acronym: NISIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: UF9467; 2014-A01313-44 (Other: ANSM)
Record Dates: First submitted 2016-06-30; First posted 2016-07-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-06

CONDITIONS: Major Depressive Episode; Suicidal Behavior
Keywords: Psychiatry; Depressive disorder; Suicide; Inflammation
MeSH Terms: conditions — Depressive Disorder; Suicide; Inflammation | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Depressive patients (Other): Blood samples (inflammatory biomarkers and genetic purpose) on depressive patients with or without story of suicidal behavior
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — Blood sample in order to study inflammatory biomarkers and genetics purpose

SUMMARY:
Suicide is a major health problem that causes annually a million death worlwide. In the stress-vulnerability model, suicidal behavior (SB) results from the interaction between an individual's predisposition (personality, family history of SB…) and stressful conditions (early life adversity).

Studies show that suicide ideations could favour inflammation and that depression is associated with an elevated inflammation.

Recent evidences also suggest that inflammatory mediators play a critical role in SB.

The aim of the study is to evaluate the inflammatory markers rate on depressed patients with or without personal history of SB.

In the second part of the study, the relations between the rates of inflammatory markers and characteristics of SB, impulsivity, psychological pain, childhood abuse and gene expression of 5HT2B receptor will be investigated.

DETAILED DESCRIPTION:
Over one year, we will recruit 280 patients suffering from a major depressive episode with (n=140) and without any history of suicide attempt (n=140), from a specialized clinic for mood disorders and SB.

First visit : clinical, biological and neuropsychological assessment

Second visit, at 6 month : Follow-up visit in the department or interview by telephone in order to assess suicidal ideations or suicide attempts since the inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Ages of 18 and 65
* Main diagnosis of major depressive episode (DSM-IV criteria)
* Having signed the informed consent
* Able to understand nature, aims, and methodology of the study

Specifics Inclusion criteria:

* Depressed patients with suicide attempt history :

  * Have done in his lifetime at least one suicide attempt (however the period of time between inclusion and suicide attempt)
* Depressed patients without suicide attempt history :

  * Had never realized suicide attempt in his lifetime

Exclusion Criteria:

* Patients suffering from inflammatories pathology
* Antibiotic or anti-inflammatory current treatment
* Pregnancy
* Participation in another clinical trial with an exclusion period
* Patient on protective measures (guardianship or trusteeship)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-05 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Rate of interleukin 2 (Il2) in a blood sample | inclusion visit
  Comparison of Il2 levels between patients with and without suicidal behaviour

SECONDARY OUTCOMES:
Rate of inflammation markers (Interleukin 1, 4, 6, 8, 10, Tumor necrosis factor alpha (TNF-a), Interferon gamma (IFNg), Vascular endothelial growth factor (VEGF), kynurenin and c-reactive protein (CRP) in a blood sample | inclusion visit
  Comparison of the levels of theses markers between patients with and without suicidal behaviour
Rate of inflammation markers and suicide attempt | inclusion visit
  Comparison of rate bloodmarkers inflammation (Il1, 4, 6, 8, 10, TNF-a, IFNg, VEGF, kynurenine and CRP) in depressed patients with latest suicide attempt and depressed patients with an history of suicide attempt
Rate of inflammation markers and violent suicide attempt | inclusion visit
  Comparison of rate bloodmarkers inflammation (Il1, 4, 6, 8, 10, TNF-a, IFNg, VEGF, kynurenine and CRP) in depressed patients with and without violent suicide attempt
Rate of inflammation markers and suicide ideations | inclusion visit
  Comparison of rate bloddmarkers (Il1, 4, 6, 8, 10, TNF-a, IFNg, VEGF, kynurenine and CRP) in depressed patients with and without current suicide ideation
Relation between markers of inflammation and suicidal behavior characteristics | inclusion visit
  Studying relations with bloodmarkers inflammation rate (Il1, 4, 6, 8, 10, TNF-a, IFNg, VEGF, kynurenine and CRP) and suicidal behaviour characteristics (the last and the most serious) (intentionality, planification, lethality)
Relation between markers of inflammation and impulsivity | inclusion visit
  Studying relations with bloodmarkers inflammation rate (Il1, 4, 6, 8, 10, TNF-a, IFNg, VEGF, kynurenine and CRP) and impulsivity (by Baratt Impulsivity Scale and neuropsychological tests)
Relation between markers of inflammation and psychological pain | inclusion visit
  Studying relations with bloodmarkers inflammation rate (Il1, 4, 6, 8, 10, TNF-a, IFNg, VEGF, kynurenine and CRP) and psychological pain (by Likert scale)
Relation between markers of inflammation and child abuse | inclusion visit
  Studying relations with bloodmarkers inflammation rate (Il1, 4, 6, 8, 10, TNF-a, IFNg, VEGF, kynurenine and CRP) and child abuse
Relation between markers of inflammation and gene expression | inclusion visit
  Studying relations with bloodmarkers inflammation rate (Il1, 4, 6, 8, 10, TNF-a, IFNg, VEGF, kynurenine and CRP) and gene expression of 5HT2B receptor
Markers of inflammation as a risk factor for suicidal behavior | at 6 months
  Studying bloodmarkers inflammation rate (Il1, 4, 6, 8, 10, TNF-a, IFNg, VEGF, kynurenine and CRP) as suicidal behaviour risk factor (suicide ideations and/or suicide attempt) with a 6 months follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No